CLINICAL TRIAL: NCT05310773
Title: Multilevel Strategies & Tailored HIV Prevention and Care for Young Couples Who Use Alcohol and Other Drugs Across Cape Town: Couples Health CoOp Plus
Brief Title: Couples Health CoOp Plus
Acronym: CHC+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, Felicia A. Browne, ScD, MPH, Senior Research Social Epidemiologist, RTI International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R01DA049612 (NIH)
Record Dates: First submitted 2022-02-21; First posted 2022-04-05 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: HIV; Substance Use; Stigma, Social
Keywords: Pre-exposure prophylaxis (PrEP); Antiretroviral therapy (ART); Alcohol and other drugs (AODs); Human Immunodeficiency Virus (HIV); Couples; Substance use; Stigma; Couples Health CoOp (CHC); South Africa; Undetectable=Untransmittable (U=U); Status-neutral
MeSH Terms: conditions — Substance-Related Disorders; Social Stigma; Acquired Immunodeficiency Syndrome | interventions — Clathrin Heavy Chains

STUDY DESIGN:
Intervention Model Description: 24 communities in clinic catchment areas (clinics selected and approved by City Health) that provide antiretroviral therapy (ART) and pre-exposure prophylaxis (PrEP) were randomly assigned to the four arms of the study (6 communities per arm). Arm 1 received the stigma awareness and education workshop and HIV testing services (HTS)/pre-exposure prophylaxis (PrEP)/anti-retroviral therapy (ART) but no Couples Health CoOp Plus (CHC+); Arm 2 received the stigma awareness and education workshop with HTS/PrEP/ART and CHC+; Arm 3 received neither the stigma awareness and education workshop nor CHC+ but received HTS/PrEP/ART; and Arm 4 received HTS/PrEP/ART and CHC+ but not the stigma awareness and education workshop. All communities received the community stigma assessments at baseline, 4 months, and 8 months follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Community Stigma Awareness and Education Workshop and HTS/ART/PrEP Only (Experimental): Communities/catchment areas randomized to this arm completed the community stigma assessments and received the community stigma awareness and education workshops. Couples had access to standard HIV testing services (HTS) with antiretroviral therapy (ART)/pre-exposure prophylaxis (PrEP) but not the Couples Health CoOp Plus (CHC+) intervention.
  Interventions: Behavioral: Community Stigma Awareness and Education Workshop
- Community Stigma Awareness and Education Workshop and HTS/ART/PrEP with CHC+ (Experimental): Communities/catchment areas randomized to this arm completed the community stigma assessments and received the community stigma awareness and education workshops. Couples had access to the Couples Health CoOp Plus (CHC+) intervention and standard HTS with antiretroviral therapy (ART)/pre-exposure prophylaxis (PrEP).
  Interventions: Behavioral: Community Stigma Awareness and Education Workshop; Behavioral: Couples Health CoOp Plus (CHC+)
- No Community Stigma Awareness and Education Workshop and HTS/ART/PrEP Only (No Intervention): Communities/catchment areas randomized to this arm completed the community stigma assessments but did not receive the community stigma awareness and education workshops. Couples had access to standard HIV testing services (HTS) with antiretroviral therapy (ART)/pre-exposure prophylaxis (PrEP) but not the Couples Health CoOp Plus (CHC+) intervention.
- No Community Stigma Awareness and Education Workshop and HTS/ART/PrEP with CHC+ (Experimental): Communities/catchment areas randomized to this arm completed the community assessments but not the community stigma awareness and education workshops. Couples had access to the Couples Health CoOp Plus (CHC+) intervention and standard HIV testing services (HTS) with antiretroviral therapy (ART)/pre-exposure prophylaxis (PrEP).
  Interventions: Behavioral: Couples Health CoOp Plus (CHC+)

INTERVENTIONS:
Behavioral: Community Stigma Awareness and Education Workshop — Key aspects of the workshop included community stigma awareness of people living with HIV, use of antiretroviral therapy (ART), pre-exposure prophylaxis (PrEP) for prevention of HIV and attitudes towards people who use alcohol and drugs. The workshop adapted a stigma-reduction curriculum based on a stigma-reduction toolkit and community HIV prevention project with community peers with skits to address stigmatizing attitudes and behaviors toward young women and men who use AODs and who may need health services, including HIV treatment and prevention. Selected modules were modified from the existing clinic-based training to fit community stigma awareness and attitudes to focus on aspects of stigma specific to young women and men who engage in syndemic-related behaviors who live in their communities. The stigma awareness and education workshop was delivered in communities randomized to receive workshops (N=12 communities).
  Arms: Community Stigma Awareness and Education Workshop and HTS/ART/PrEP Only; Community Stigma Awareness and Education Workshop and HTS/ART/PrEP with CHC+
Behavioral: Couples Health CoOp Plus (CHC+) — The Couples Health CoOp Plus (CHC+) was adapted from the initial Couples Health CoOp (CHC)-an empowerment-based intervention developed for South African couples that addresses the syndemic of alcohol and other drug (AOD) use, violence, and HIV risk. It is grounded in Social Cognitive Theory and promotes prevention strategies that address the relational context of equality in which sexual risk takes place. The adapted Couples Health CoOp Plus (CHC+) incorporated antiretroviral therapy (ART)/pre-exposure prophylaxis (PrEP) for a biobehavioral approach with an emphasis on uptake and good adherence (N=12 communities; N=240 couples).
  Arms: Community Stigma Awareness and Education Workshop and HTS/ART/PrEP with CHC+; No Community Stigma Awareness and Education Workshop and HTS/ART/PrEP with CHC+

SUMMARY:
This study addresses HIV prevention and treatment for young couples living in Cape Town, South Africa, through a comprehensive biobehavioral multilevel approach-the Couples Health CoOp Plus (CHC+).

Through a cluster randomized trial with a modified factorial design, 24 Cape Town communities consisting of catchment areas for clinics that provide antiretroviral therapy (ART) and pre-exposure prophylaxis (PrEP), received either a stigma awareness and education workshop or no workshop with repeated measures. Within clinic catchment areas, 481 couples (young women and their primary male sex partners both aged 18 to 30) were recruited. These couples received HIV testing services (HTS) and/or the Couples Health CoOp Plus (CHC+), depending on their intervention arm.

The overarching aim of these interventions is to prevent new cases of HIV. It is hypothesized that communities that are assigned to the stigma awareness and education workshop will demonstrate higher levels of social acceptance and fewer cases of enacted/experienced stigma at the community level. Additionally, it is expected couples assigned to the Couples Health CoOp Plus (CHC+) intervention will have greater antiretroviral therapy (ART)/pre-exposure prophylaxis (PrEP) initiation and adherence, lower alcohol and other drug (AOD) use, less sexual risk, less violence, and more positive relationship norms and communication.

Specifically, the study aims to:

Aim 1: Modify the Couples Health CoOp (CHC) intervention to include antiretroviral therapy (ART)/pre-exposure prophylaxis (PrEP) in a formative phase and with review from the Community Collaborative Board (CCB) and Peer Advisory Board (PAB).

Aim 2: Evaluate the impact of a stigma awareness and education workshop on community members' attitudes and behaviors toward young women and men who use AODs and other people seeking HIV services (testing/ART/PrEP) and other health services at 4- and 8-month follow-up.

Aim 3: Test the efficacy of the Couples Health CoOp Plus (CHC+) to increase both partners' antiretroviral therapy (ART)/pre-exposure prophylaxis (PrEP) initiation and adherence (primary outcome) and reduce alcohol and other drug (AOD) use, sexual risk and violence, and enhance positive relationship norms and communication relative to HIV testing services (HTS) (secondary outcomes).

Aim 4: Examine through mixed methods the interaction of a stigma awareness and education workshop and the Couples Health CoOp Plus (CHC+) on increased antiretroviral therapy (ART)/pre-exposure prophylaxis (PrEP) and initiation, retention, and adherence among young women and their primary partners.

DETAILED DESCRIPTION:
The Couples Health CoOp Plus (CHC+) was adapted from the Couples Health CoOp (CHC)-an empowerment-based intervention developed for South African couples that addresses the syndemic of alcohol and other drug (AOD) use, violence, and HIV risk. It is grounded in Social Cognitive Theory and promoted prevention strategies that addressed the relational context of equality in which sexual risk takes place. The Couples Health CoOp (CHC) has demonstrated efficacy in increasing condom use, improving relationship norms, decreasing heavy alcohol use among men, and decreasing HIV incidence among women. Long-term benefits of the Couples Health CoOp (CHC) have been explored including women reporting less fighting with their partner and men reporting being more faithful and loving. As part of this current study (Aim 1), the behavioral Couples Health CoOp (CHC) was adapted to include biomedical HIV strategies antiretroviral therapy (ART)/pre-exposure prophylaxis (PrEP) and updated materials. Formative qualitative work with a Community Collaborative Board (CCB) and a Peer Advisory Board (PAB) guided the adaptation and updating of the Couples Health CoOp Plus (CHC+) intervention. The Couples Health CoOp Plus (CHC+) is a 2-module workshop delivered over two days and contains didactic and experiential lessons on alcohol and other drug (AOD) use, a status-neutral approach to the prevention and management of HIV, sexual and reproductive health (SRH), relationship norms, violence, and tools to improve communication.

Formative findings regarding clinic-level stigma and discrimination showed that stigma reduction training provided in communities surrounding healthcare clinics may reduce stigmatizing behaviors and attitudes that are enacted by family, friends, and other community members toward those seeking healthcare. The stigma reduction survey and workshop were developed and adapted as part of Aim 1 formative activities.

The study enrolled approximately 20 couples in each of the 24 communities in and around Cape Town, South Africa. Communities surrounding healthcare clinics were paired according to community demographic and socioeconomic factors and randomized to one of four arms:

1. stigma awareness and education workshop (community) and HIV testing services (HTS)/antiretroviral therapy (ART)/pre-exposure prophylaxis (PrEP) (couple);
2. stigma awareness and education workshop (community), and HIV testing services (HTS)/antiretroviral therapy (ART)/pre-exposure prophylaxis (PrEP) with Couples Health CoOp Plus (CHC+) (couple);
3. no stigma awareness and education workshop (community) and HIV testing services (HTS)/antiretroviral therapy (ART)/pre-exposure prophylaxis (PrEP) (couple);
4. no stigma awareness and education workshop (community), and HIV testing services (HTS)/antiretroviral therapy (ART)/pre-exposure prophylaxis (PrEP) with Couples Health CoOp Plus (CHC+) (couple).

As noted, couples in communities that were not assigned to receive the CHC+ intervention received HIV testing services (HTS), including provision of antiretroviral therapy (ART) and pre-exposure prophylaxis (PrEP) as part of standard of care.

HIV, alcohol and other drug (AOD), and pregnancy testing was conducted at baseline and at 3- and 6-month follow-up.

Assessment of community stigma occurred at baseline with all 24 communities and the stigma awareness and education workshop occurred in only those randomized to it. The follow-up occurred within all communities at 4- and 8-months post-baseline.

ELIGIBILITY:
Selected Inclusion Criteria (for Couples):

* 18 to 30 years old
* Is in a relationship with a primary partner
* Had recent condomless sex with their primary partner
* Has not taken PrEP or ART in the past 90 days
* Has drunk alcohol and/or used drugs at least once a week over the past 90 days

Selected Exclusion Criteria (for Couples):

* Not currently pregnant (for women)
* Not currently being treated for drug-resistant tuberculosis (TB)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 962 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Antiretroviral Therapy (ART) Initiation [individual and couple-level] | 3-month follow-up
  ART initiation will be measured using initiation information recorded in the participant's clinic medical record.
Antiretroviral Therapy (ART) Initiation [individual and couple-level] | 6-month follow-up
  ART initiation will be measured using initiation information recorded in the participant's clinic medical record.
Pre-Exposure Prophylaxis (PrEP) Initiation [individual and couple-level] | 3-month follow-up
  Pre-exposure prophylaxis (PrEP) initiation will be measured using initiation information recorded in the participant's clinic medical record.
Pre-Exposure Prophylaxis (PrEP) Initiation [individual and couple-level] | 6-month follow-up
  Pre-exposure prophylaxis (PrEP) initiation will be measured using initiation information recorded in the participant's clinic medical record.
Biological: Antiretroviral Therapy (ART) Adherence [individual and couple-level] | 3-month follow-up
  ART adherence will be measured using viral load or cluster of differentiation 4 (CD4) count measures recorded in the participant's medical record. Threshold for adherence will be cluster of differentiation 4 (CD4) count (more than 200) and HIV viral load (less than 50 copies per ml).
Biological: Antiretroviral Therapy (ART) Adherence [individual and couple-level] | 6-month follow-up
  ART adherence will be measured using viral load or cluster of differentiation 4 (CD4) count measures recorded in the participant's medical record. Threshold for adherence will be cluster of differentiation 4 (CD4) count (more than 200) and HIV viral load (less than 50 copies per ml).
Self-Report: Antiretroviral Therapy (ART) Adherence [individual and couple-level] | 3-month follow-up
  Self-report past 30-day use, missed doses and patterns of use of antiretroviral therapy (ART) for self-report adherence will be measured using the Revised Risk Behavior Assessment (RRBA)/Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Antiretroviral Therapy (ART) Adherence [individual and couple-level] | 6-month follow-up
  Self-report past 30-day use, missed doses and patterns of use of antiretroviral therapy (ART) for self-report adherence will be measured using the Revised Risk Behavior Assessment (RRBA)/Pretoria Risk Behavior Assessment (PRBA+).
Biological: Pre-Exposure Prophylaxis (PrEP) Adherence [individual and couple-level] | 3-month follow-up
  Tenofovir Diphosphate (TFV-DP) and FTC Triphosphate (FTC-TP) concentrations in dried blood spots (DBS) with drug concentrations of greater than 700 femtomoles (fmol)/liters(L) will be considered adherent to pre-exposure prophylaxis (PrEP).
Biological: Pre-Exposure Prophylaxis (PrEP) Adherence [individual and couple-level] | 6-month follow-up
  Tenofovir Diphosphate (TFV-DP) and FTC Triphosphate (FTC-TP) concentrations in dried blood spots (DBS) with drug concentrations of greater than 700 femtomoles (fmol)/liters(L) will be considered adherent to pre-exposure prophylaxis (PrEP).
Self-Report: Pre-Exposure Prophylaxis (PrEP) Adherence [individual and couple-level] | 3-month follow-up
  Self-report past 30-day use, missed doses and patterns of use of pre-exposure prophylaxis (PrEP) for self-report adherence will be measured using the Revised Risk Behavior Assessment (RRBA)/Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Pre-Exposure Prophylaxis (PrEP) Adherence [individual and couple-level] | 6-month follow-up
  Self-report past 30-day use, missed doses and patterns of use of pre-exposure prophylaxis (PrEP) for self-report adherence will be measured using the Revised Risk Behavior Assessment (RRBA)/Pretoria Risk Behavior Assessment (PRBA+).
Antiretroviral Therapy (ART) Persistence and Discontinuation [individual and couple-level] | 3-month follow-up
  Number of antiretroviral therapy (ART) refills since initiation recorded in clinic medical records.
Antiretroviral Therapy (ART) Persistence and Discontinuation [individual and couple-level] | 6-month follow-up
  Number of antiretroviral therapy (ART) refills since initiation recorded in clinic medical records.
Self-Report: Antiretroviral therapy (ART) Persistence and Discontinuation [individual and couple-level] | 3-month follow-up
  Self-reported time in months on antiretroviral therapy (ART) since initiation will be measured using the Revised Risk Behavior Assessment (RRBA)/Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Antiretroviral therapy (ART) Persistence and Discontinuation [individual and couple-level] | 6-month follow-up
  Self-reported time in months on antiretroviral therapy (ART) since initiation will be measured using the Revised Risk Behavior Assessment (RRBA)/Pretoria Risk Behavior Assessment (PRBA+).
Data Extraction: Pre-Exposure Prophylaxis (PrEP) Persistence and Discontinuation [individual and couple-level | 3-month follow-up
  Number of pre-exposure prophylaxis (PrEP) refills since initiation as recorded clinic medical records.
Data Extraction: Pre-Exposure Prophylaxis (PrEP) Persistence and Discontinuation [individual and couple-level | 6-month follow-up
  Number of pre-exposure prophylaxis (PrEP) refills since initiation as recorded clinic medical records.
Self-Report: Pre-Exposure Prophylaxis (PrEP) Persistence and Discontinuation [individual and couple-level] | 3-month follow-up
  Self-reported time in months on pre-exposure prophylaxis (PrEP) since initiation on pre-exposure prophylaxis (PrEP) will be measured using the Revised Risk Behavior Assessment (RRBA)/Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Pre-Exposure Prophylaxis (PrEP) Persistence and Discontinuation [individual and couple-level] | 6-month follow-up
  Self-reported time in months on pre-exposure prophylaxis (PrEP) since initiation on pre-exposure prophylaxis (PrEP) will be measured using the Revised Risk Behavior Assessment (RRBA)/Pretoria Risk Behavior Assessment (PRBA+).
Data Extraction: Antiretroviral therapy (ART) Retention | 3-month follow-up
  Antiretroviral therapy (ART) retention in care will be measured as attendance to follow-up visits as recorded in clinic medical records.
Data Extraction: Antiretroviral therapy (ART) Retention | 6-month follow-up
  Antiretroviral therapy (ART) retention in care will be measured as attendance to follow-up visits as recorded in clinic medical records.
Self-Report: Pre-exposure Prophylaxis (PrEP) Retention [individual and couple-level] | 3-month follow-up
  Self-report pre-exposure prophylaxis (PrEP) retention in care will be measured as attendance to follow-up visits using the Revised Risk Behavior Assessment (RRBA)/Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Pre-exposure Prophylaxis (PrEP) Retention [individual and couple-level] | 6-month follow-up
  Self-report pre-exposure prophylaxis (PrEP) retention in care will be measured as attendance to follow-up visits using the Revised Risk Behavior Assessment (RRBA)/Pretoria Risk Behavior Assessment (PRBA+).

SECONDARY OUTCOMES:
Community Stigma [structural level] | Baseline
  Surveys will be used to measure stigmatizing attitudes and perceptions towards people who use alcohol and other drugs (AODs), living with HIV and seeking and antiretroviral therapy (ART) or pre-exposure prophylaxis (PrEP) services for prevention. Greater values indicate higher levels of community-level stigma and discrimination.
Community Stigma [structural level] | 4-month follow-up
  Surveys will be used to measure stigmatizing attitudes and perceptions towards people who use alcohol and other drugs (AODs), living with HIV and seeking and antiretroviral therapy (ART) or pre-exposure prophylaxis (PrEP) services for prevention. Greater values indicate higher levels of community-level stigma and discrimination.
Community Stigma [structural level] | 8-month follow-up
  Surveys will be used to measure stigmatizing attitudes and perceptions towards people who use alcohol and other drugs (AODs), living with HIV and seeking and antiretroviral therapy (ART) or pre-exposure prophylaxis (PrEP) services for prevention. Greater values indicate higher levels of community-level stigma and discrimination.
Biological: Drug use [individual level] | Baseline
  Recent drug use (amphetamine, cocaine, methamphetamine, marijuana [THC], opiates and/or Mandrax) will be measured using a rapid urine-based drug screening test panel.
Biological: Drug use [individual level] | 3-month follow-up
  Recent drug use (amphetamine, cocaine, methamphetamine, marijuana [THC], opiates and/or Mandrax) will be measured using a rapid urine-based drug screening test panel.
Biological: Drug use [individual level] | 6-month follow-up
  Recent drug use (amphetamine, cocaine, methamphetamine, marijuana [THC], opiates and/or Mandrax) will be measured using a rapid urine-based drug screening test panel.
Biological: Alcohol use [individual level] | Baseline
  Recent alcohol (last 10 days) use will be measured by the presence of ethyl glucuronide (EtG), a breakdown product of ethanol, using an ethyl glucuronide (EtG) urine test.
Biological: Alcohol use [individual level] | 3-month follow-up
  Recent alcohol (last 10 days) use will be measured by the presence of ethyl glucuronide (EtG), a breakdown product of ethanol, using an ethyl glucuronide (EtG) urine test.
Biological: Alcohol use [individual level] | 6-month follow-up
  Recent alcohol (last 10 days) use will be measured by the presence of ethyl glucuronide (EtG), a breakdown product of ethanol, using an ethyl glucuronide (EtG) urine test.
Self-Report: Violence [individual and couple-level] | Baseline
  Self-report emotional, physical, and sexual abuse, recent victimization, and family violence & experience of physical & sexual abuse will be measured using the World Health Organization (WHO) assessment of emotional, physical, & sexual abuse and the Revised Risk Behavior Assessment (RRBA).
Self-Report: Violence [individual and couple-level] | 3-month follow-up
  Self-report emotional, physical, and sexual abuse, recent victimization, and family violence & experience of physical & sexual abuse will be measured using the World Health Organization (WHO) assessment of emotional, physical, & sexual abuse and the Revised Risk Behavior Assessment (RRBA).
Self-Report: Violence [individual and couple-level] | 6-month follow-up
  Self-report emotional, physical, and sexual abuse, recent victimization, and family violence & experience of physical & sexual abuse will be measured using the World Health Organization (WHO) assessment of emotional, physical, & sexual abuse and the Revised Risk Behavior Assessment (RRBA).
Self-Report: Sexual Risk [individual and couple-level] | Baseline
  Self-reported frequency of condom use at last sex over the past 3 months measured by the Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Sexual Risk [individual and couple-level] | 3-month follow-up
  Self-reported frequency of condom use at last sex over the past 3 months measured by the Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Sexual Risk [individual and couple-level] | 6-month follow-up
  Self-reported frequency of condom use at last sex over the past 3 months measured by the Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Sexual Risk [individual and couple-level] | Baseline
  Self-reported frequency of alcohol and other drug (AOD) use prior to sex in the last 3 months as measured by the Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Sexual Risk [individual and couple-level] | 3-month follow-up
  Self-reported frequency of alcohol and other drug (AOD) use prior to sex in the last 3 months as measured by the Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Sexual Risk [individual and couple-level] | 6-month follow-up
  Self-reported frequency of alcohol and other drug (AOD) use prior to sex in the last 3 months as measured by the Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Sexual Risk [individual and couple-level] | Baseline
  Self-reported number of sex partners, concurrent sexual partners and sex trading partners over the past 3 months measured by the Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Sexual Risk [individual and couple-level] | 3-month follow-up
  Self-reported number of sex partners, concurrent sexual partners and sex trading partners over the past 3 months measured by the Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Sexual Risk [individual and couple-level] | 6-month follow-up
  Self-reported number of sex partners, concurrent sexual partners and sex trading partners over the past 3 months measured by the Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Sexual Risk [individual and couple-level] | Baseline
  Self-report responses on the single item measured by the Pretoria Risk Behavior Assessment (PRBA+) will be used to assess use of contraception and types of contraception.
Self-Report: Sexual Risk [individual and couple-level] | 3-month follow-up
  Self-report responses on the single item measured by the Pretoria Risk Behavior Assessment (PRBA+) will be used to assess use of contraception and types of contraception.
Self-Report: Sexual Risk [individual and couple-level] | 6-month follow-up
  Self-report responses on the single item measured by the Pretoria Risk Behavior Assessment (PRBA+) will be used to assess use of contraception and types of contraception.
Self-Report: Relationship Norms [individual and couple-level] | Baseline
  Self-reported attitudes about traditional relationship roles, empowerment, and assertiveness will be measured by a modified scale assessing beliefs about relationship norms and the Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Relationship Norms [individual and couple-level] | 3-month follow-up
  Self-reported attitudes about traditional relationship roles, empowerment, and assertiveness will be measured by a modified scale assessing beliefs about relationship norms and the Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Relationship Norms [individual and couple-level] | 6-month follow-up
  Self-reported attitudes about traditional relationship roles, empowerment, and assertiveness will be measured by a modified scale assessing beliefs about relationship norms and the Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Communication [individual and couple-level] | Baseline
  Self-reported communication between partners regarding testing, HIV and sexually transmitted infection (STI) status, other partners, sexual negotiation, and condom use as measured by the Revised Risk Behavior Assessment (RRBA)/Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Communication [individual and couple-level] | 3-month follow-up
  Self-reported communication between partners regarding testing, HIV and sexually transmitted infection (STI) status, other partners, sexual negotiation, and condom use as measured by the Revised Risk Behavior Assessment (RRBA)/Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Communication [individual and couple-level] | 6-month follow-up
  Self-reported communication between partners regarding testing, HIV and sexually transmitted infection (STI) status, other partners, sexual negotiation, and condom use as measured by the Revised Risk Behavior Assessment (RRBA)/Pretoria Risk Behavior Assessment (PRBA+).
Self-Report: Observed or Knowledge of Stigma [individual and couple-level] | Baseline
  Observations or knowledge of stigma perpetrated by others in the community will be measured by stigma items adapted from previous research.
Self-Report: Observed or Knowledge of Stigma [individual and couple-level] | 3-month follow-up
  Observations or knowledge of stigma perpetrated by others in the community will be measured by stigma items adapted from previous research.
Self-Report: Observed or Knowledge of Stigma [individual and couple-level] | 6-month follow-up
  Observations or knowledge of stigma perpetrated by others in the community will be measured by stigma items adapted from previous research.

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Browne, ScD, MPH, Principal Investigator — RTI International; Tara Carney, PhD, Principal Investigator — Medical Research Council, South Africa
Locations (1):
- South African Medical Research Council, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wechsberg WM, Carney T, Browne FA, van der Drift IM, Kline TL, Nyblade LL, Ndirangu J, Orrell C, Bonner CP, Caron E. Multilevel strategies to end HIV for young couples in Cape Town: Study protocol for a cluster randomized trial. PLoS One. 2024 Jun 7;19(6):e0305056. doi: 10.1371/journal.pone.0305056. eCollection 2024. PMID 38848400